CLINICAL TRIAL: NCT05494463
Title: Comparison of the Miller Laryngoscope and the Macintosh Laryngoscope During Endotracheal Intubation in Adult Patients
Brief Title: Miller Blade for Intubation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RNN/103/22/KE
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2022-07

CONDITIONS: Intubation Complication
Keywords: laryngoscopy; endotracheal intubation; Miller blade; Macintosh blade

STUDY DESIGN:
Intervention Model Description: First laryngoscopy with randomly choosed blade and then laryngoscopy wiht second choosen blade in the same patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Macintosh blade (No Intervention): laryngoscopy with Macintosh blade
- Miller blade (Active Comparator): laryngoscopy with Miller blade in the same patient
  Interventions: Device: Miller blade

INTERVENTIONS:
Device: Miller blade — After laryngoscopy with Macintosh blade patient will be evaluated in laryngoscopy with Miller blade
  Arms: Miller blade

SUMMARY:
The study compares laryngeal view obtained with standard Macintosh blade laryngoscope and Miller blade laryngoscope in adult patients. After introduction to general anesthesia anesthesiologist will perform laryngoscopy with one chosen blade and after evaluation of visualisation of entrance to larynx will change blade to second one and repeat evaluation.

DETAILED DESCRIPTION:
Tracheal intubation is the gold standard of the airway in the operating theater in patients undergoing general anesthesia for surgery, in intensive care and emergency medicine, in patients with severe respiratory failure, which is life-threatening. The laryngoscope is a device used to visualize the entrance to the airway and the subsequent insertion of the tracheal tube into the trachea and main bronchus. Macintosh and Miller laryngoscopes have been used in clinical practice for several decades. The Macintosh laryngoscope is most commonly used for the intubation of adult patients, and the Miller laryngoscope for the intubation of newborns, including premature babies and pediatric patients. Currently, when we are dealing with the sars covid-19 virus epidemic and a large number of patients with respiratory failure requiring endotracheal intubation and replacement ventilation, searching for a device that facilitates endotracheal intubation, especially by people with little experience in using it, in the absence of anesthesiologists, seems to be justified. The aim of the study will be to assess the possibility of using the Miller's laryngoscope for intubation of adult patients and to compare it with the most frequently used Macintosh laryngoscope in this group of patients. The study will include patients scheduled for elective surgery under general endotracheal anesthesia. After a typical induction of anesthesia with the use of short-term intravenous anesthetics, opioids and muscle relaxants, appropriate for the planned surgery and a specific patient, after obtaining complete neuromuscular blockade, a Macintosh laryngoscope will be inserted to perform direct laryngoscopy and assess the exit to the respiratory tract with the help of the Cormack scale. Then the laryngoscope will be removed, the patient will receive active oxygen therapy to increase blood oxygenation to the value of 99-100%, and then an additional dose of intravenous anesthetic will be administered and a second direct laryngoscopy will be performed with the Miller's laryngoscope with a subsequent assessment of airway entry using the scale Cormack. The patient will then be intubated and connected to an anesthesia machine.

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for elective procedures under general anesthesia with endotracheal intubation

Exclusion Criteria:

* patients with expected difficutl intubation requiring advanced intubation techniques
* with injuries of the cervical spine, or for surgery in the cervical spine
* patients with increased intracranial and intraocular pressure, with vascular changes in the CNS and other parts of the body
* patients with ASA III and above
* patients who do not consent to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1130 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Number of Grade of view of entrance to larynx | immediate
  Laryngoscopy with Macintosh blade and then with Miller blade in the same patient, grade of view estimated in Cormack-lehane scale and POGO - percentage of glottis opening

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ratajczyk P, Kluj P, Szmyd B, Resch J, Hogendorf P, Durczynski A, Gaszynski T. A Comparison of Miller Straight Blade and Macintosh Blade Laryngoscopes for Intubation in Morbidly Obese Patients. J Clin Med. 2024 Jan 24;13(3):681. doi: 10.3390/jcm13030681. PMID 38337375